CLINICAL TRIAL: NCT05872425
Title: Efficacy and Safety of Dingkundan Combined With Combination Oral Contraceptives in the Treatment of PCOS: an Open-label, Non-randomized Controlled Clinical Study
Brief Title: Efficacy and Safety of Dingkundan Combined With Combination Oral Contraceptives in the Treatment of PCOS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Guangdong Women and Children Hospital (Other)
Responsible Party: Principal Investigator, Li Li, Deputy Director, Institute of Women's and Children's Health, Guangdong Women and Children Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GuangdongWCH-LiLi
Record Dates: First submitted 2023-04-27; First posted 2023-05-24 (Actual); Last update posted 2024-05-30 (Actual); Status verified 2024-05

CONDITIONS: PCOS
Keywords: Dingkundan(DKP); Compound Oral Contraceptives(COC); PCOS
MeSH Terms: interventions — drospirenone; Ethinyl Estradiol

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Treatment with DingKunDan(GuangYuYuan) combined with compound oral contraceptives (Experimental): This arm is treated with DingKunDan plus compound oral contraceptives: Drospirenone and Ethinylestradiol Tablets (Ⅱ).
  Interventions: Drug: DingKunDan(GuangYuYuan); Drug: Drospirenone and Ethinylestradiol Tablets (Ⅱ)
- Treatment with compound oral contraceptives (Active Comparator): This arm is only treated with compound oral contraceptives: Drospirenone and Ethinylestradiol Tablets (Ⅱ).
  Interventions: Drug: DingKunDan(GuangYuYuan)

INTERVENTIONS:
Drug: DingKunDan(GuangYuYuan) — The experimental group would be given DingKunDan, the subjects should take 3.5g each time, twice a day.
  Subjects in the control group only needed to take COC. Both groups take medicine for 3 months consecutively as a course of treatment.
  Other Names: DingKunDan(GuangYuYuan): Z20059003; Drospirenone and Ethinylestradiol Tablets (Ⅱ): H20140972
Drug: Drospirenone and Ethinylestradiol Tablets (Ⅱ) — The experimental group and the control group would be given oral Drospirenone and Ethinylestradiol Tablets (Ⅱ). According to the packaging instructions, on the first day of menstruation, according to the packaging instructions, the subjects should take the tablet, then take the rest sequential at the same time every day for 28 consecutive days, menstruation would happen after drug withdrawal (or after 7 days of drug withdrawal), and the next medication cycle begin on the first day of menstruation.
  Other Names: Drospirenone and Ethinylestradiol Tablets (Ⅱ): H20140972
  Arms: Treatment with DingKunDan(GuangYuYuan) combined with compound oral contraceptives

SUMMARY:
This is a single-center, non-randomized, open-label clinical study to investigate the efficacy and safety of Dingkundan (DKP) combined with compound oral contraceptives (COC) in the treatment of PCOS. This study is mainly to compare the effect of COC plus DKP verse COC on reducing androgen, improving the function of ovarian and the individual metabolism. The secondary objective of our study is to explore the efficacy of DKP on pregnancy in patients with PCOS and its safety.

DETAILED DESCRIPTION:
In this study, the decreased level of serum androgen was used as the main outcome index. It was assumed that PCOS patients treated with Dingkundan combined with compound oral contraceptives for 3 menstrual cycles had decreased serum androgen by 0.53nmol/L. It was assumed that the serum androgen decreased by 0.21nmol/L after 3 menstrual cycles of combined oral contraceptives alone. If α = 0.05, the test degree was 80%, and the dropout rate of 20%, considering that the sample size ratio between the experimental group and control group was 1, the sample size of experimental group and control group were 60 cases each, and 120 cases in total. All the samples were recruited from the Department of Gynecology and Women's Health Care of Guangdong Women and Children's Health Hospital.

This study was approved by the Ethics Committee of the hospital, and all participants are required to sign informed consent.

Before the study, researchers should be trained in a unified and standardized manner, including medication methods, observation indicators, judgment and treatment of adverse reactions/events, and reporting of serious adverse events.

The researcher must adequately and accurately record the research process so that the research data can be verified. These records can be divided into two categories: study documents and raw patient data. Study documents include protocols and amendments, sample informed consent forms, researcher resumes and authorization forms, and other required documents and correspondence. Original documents of patients' include patient inpatient/outpatient records, doctor's and nurse's orders, appointment dates, original laboratory reports, ultrasound, signed informed consent forms, patient screening forms, etc.

During the study period, if the subject withdraws the informed consent, or refuses the further follow-up, or loses follow-up, or dies, the sample will be disqualified.

If the subject withdraws consent, refuses to continue the study, or the investigator determines that the subject's clinical symptoms/physical condition has worsened and that the subject is no longer suitable for the study, or the subject develops toxicity intolerance, such as any clinical AE, laboratory abnormalitiesor, or the investigator determines that the subject has reached the study endpoint, or any circumstances warrant discontinuation of this study judged by the investigator, or the study sponsor discontinues the study, this study will be stop.

Anyway, this clinical study is conducted in accordance with the Declaration of Helsinki and relevant regulations on clinical trials in China. It can only be carried out after obtaining the approval of the Ethics Committee. The modification of clinical research protocols, informed documents and other materials involved in clinical research should be approved by the Ethics Committee before implementation. The investigator should protect the rights and privacy of the subject.

ELIGIBILITY:
Inclusion Criteria:

* Women diagnosed with PCOS.
* Aged from 18 to 35 years old, in the reproductive age.
* Have not taken any hormone or Chinese medicine in the past 3 months.

Exclusion Criteria:

* Age < 18 years or > 35 years.
* Have taken hormones or Chinese medicine in the last 3 months.
* Have congenital adrenal hyperplasia, Cushing's syndrome, or androgen-secreting tumors.
* Abnormal function of liver and kidney.
* Have hrombotic disease, arterial or venous thromboembolism, or major organic disease.

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — Female
Enrollment: 120 (Actual)
Dates: Start 2023-02-01 (Actual); Primary Completion 2024-04-01 (Actual); Study Completion 2024-04-01 (Actual)

PRIMARY OUTCOMES:
Serum androgen | Before inclusion；after one treatment course.
  Basic serum androgen is one of the primary outcome measure and is aim to evaluate the efficacy of Dingkundan that as an adjuvant therapy for PCOS.
Free testosterone | Before inclusion；after one treatment course.
  Free testosterones is one of the primary outcome measureis aim to evaluate the efficacy of Dingkundan that as an adjuvant therapy for PCOS.
Androstenedione | Before inclusion；after one treatment course.
  Androstenedione is one of the primary outcome measure is aim to evaluate the efficacy of Dingkundan that as an adjuvant therapy for PCOS.
sex hormone-binding globulin（SHBG） | Before inclusion；after one treatment course.
  SHBG is one of the primary outcome measure is aim to evaluate the efficacy of Dingkundan that as an adjuvant therapy for PCOS.

SECONDARY OUTCOMES:
Fasting blood-glucose (FBG) | Before inclusion；after one treatment course.
  This outcome measure is aim to assess if Dingkundan is a useful adjuvant therapy for PCOS in improving metabolism.
Fasting insulin (FINS) | Before inclusion；after one treatment course.
  This outcome measure is aim to assess if Dingkundan is a useful adjuvant therapy for PCOS in improving metabolism.
HOMA-IR | Before inclusion；after one treatment course.
  HOMA-IR is used to assess the level of insulin resistance and help to evaluate the metabolism of individuals.
Anti-Müllerian hormone (AMH) | Before inclusion；after one treatment course.
  AMH is an important index to evaluate AMH is an important index to evaluate the reserve function of ovarian.
HCY | Before inclusion；after one treatment course.
  HCY is used to assess the level of folate metabolism

OTHER OUTCOMES:
Adverse reaction | 3 months after one treatment course.
  Adverse reaction is used to assess the safety level of DingKunDan. Adverse reactions were reported by the patient, such as nausea, vomiting, decreased appetite, irregular uterine bleeding, and breast tenderness.
Liver function | 3 months after one treatment course.
  Liver function is used to assess the safety level of DingKunDan. Liver function includes the level of ALT, AST, ALT/AST by blood test.
Kidney function | 3 months after one treatment course.
  Kidney function is used to assess the safety level of DingKunDan. Kidney function includes the level of Urea, CO2, CRE, UA, β2-MG by blood test.

CONTACTS AND LOCATIONS:
Locations (1):
- Guangdong Women and Children Health Hospital, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: Undecided

DOCUMENTS (2):
  • Study Protocol (2023-02-01): https://cdn.clinicaltrials.gov/large-docs/25/NCT05872425/Prot_000.pdf
  • Informed Consent Form (2023-02-01): https://cdn.clinicaltrials.gov/large-docs/25/NCT05872425/ICF_001.pdf